CLINICAL TRIAL: NCT05888012
Title: Efficacy and Safety Comparison of Balloon Catheter and Basket Catheter for Endoscopic Pancreatic Duct Stone Clearance
Brief Title: Balloon Catheter vs. Basket Catheter in Pancreatic Duct Stone Clearance
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Principal Investigator, Changhai Hospital
Other Study IDs: Basket vs. Balloon
Record Dates: First submitted 2023-05-07; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pancreatitis
Keywords: Pancreatic stone; Endoscopic retrograde cholangiopancreatography (ERCP); Basket catheter; Balloon catheter; Stone clearance
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: basket catheter — Stone extraction is completed with either a basket or balloon catheter at the time of ERCP. The basket catheter is made of nickel-titanium wires which can be manipulated to trap and withdraw stones.
Device: balloon catheter — Stone extraction is completed with either a basket or balloon catheter at the time of ERCP. The balloon catheter is made of latex, which is inflated after passing the stone, thus pushing the stone outwards.

SUMMARY:
The aim of the study is to compare the safety and efficacy of the basket catheter with that of the balloon catheter for endoscopic extraction of pancreatic stones.

DETAILED DESCRIPTION:
This is a retrospective cohort study. Patients with chronic pancreatitis who underwent ERCP for pancreatic duct stone extraction using either a basket or a balloon catheter were enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* CP patients with main pancreatic duct (MPD) stones who underwent ERCP

Exclusion Criteria:

* Patients had undergone pancreatic surgery or gastrectomy with Billroth II reconstruction prior to the ERCP procedure
* Patients were suspected of having a malignant tumor
* Patients combined with bile duct stones
* Patients had severe pancreatic duct structure
* Patients with insufficient clinical data
* Patients with previous ERCP treatment
* Patients had received both catheters

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CP patients with pancreatic duct stones who underwent ERCP between February 2012 and December 2021were identified. The diagnosis of CP was established based on computed tomography, magnetic resonance imaging or endoscopic ultrasound examinations.
Sampling Method: Non-Probability Sample
Enrollment: 6493 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
the rate of stone clearance in basket and balloon catheter groups | 1 year after ERCP
  complete clearance, defined as fragmentation of the pancreatic stones to < 3 mm and clearance of more than 90% of the fragments; partial clearance, defined as clearance of 50-90% of the fragments; and unsuccessful clearance, defined as the presence of pancreatic stones ≥ 3 mm or clearance of less than 50% of the fragments.

SECONDARY OUTCOMES:
the rates of ERCP peri-procedural outcomes and the rates of complications of ERCP in basket and balloon catheter groups | 1 year after ERCP
  ERCP peri-procedural outcomes included difficult cannulation, endoscopic sphincterotomy, dilation of stenosis, and extraction through the minor papilla. Major post-ERCP complications, which were defined according to the Consensus Criteria, included post-ERCP pancreatitis (PEP), bleeding, infection, perforation, and basket impaction

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided